CLINICAL TRIAL: NCT01646177
Title: A 12-Week Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Efficacy and Safety of LY2439821 to Etanercept and Placebo in Patients With Moderate to Severe Plaque Psoriasis With a Long-Term Extension Period
Brief Title: A Study in Participants With Moderate to Severe Psoriasis (UNCOVER-3)
Acronym: UNCOVER-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13685; I1F-MC-RHBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2019-11-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept; ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo for ixekizumab administered by two SC injections at Week 0, then one SC injection per Dosing Regimen 1 until Week 12. Placebo for etanercept administered by one SC injection twice weekly starting at Week 0 up to Week 12. At Week 12, participants are assigned to Dosing Regimen 2.
  Interventions: Drug: Placebo
- 50 mg etanercept (Active Comparator): Administered by SC injections twice weekly starting at Week 0 up to Week 12. At Week 12, arm is assigned to Dosing Regimen 2
  Interventions: Drug: 50 mg etanercept
- 80 mg ixekizumab Dosing Regimen 2 (Experimental): Administered by two 80 mg SC injections at Week 0, then one 80 mg SC injection per Dosing Regimen 2 until Week 264.
  Interventions: Drug: 80 mg ixekizumab
- 80 mg ixekizumab Dosing Regimen 1 (Experimental): Administered by two 80 milligram (mg) subcutaneous (SC) injections at Week 0, then one 80 mg SC injection per Dosing Regimen 1 until Week 12. At Week 12, arm is assigned to Dosing Regimen 2.
  Interventions: Drug: 80 mg ixekizumab

INTERVENTIONS:
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: 50 mg etanercept — Administered SC
  Arms: 50 mg etanercept
Drug: 80 mg ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: 80 mg ixekizumab Dosing Regimen 1; 80 mg ixekizumab Dosing Regimen 2

SUMMARY:
This study will assess the safety and efficacy of ixekizumab (LY2439821), compared to etanercept and placebo in participants with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Presents with chronic plaque psoriasis based on a confirmed diagnosis of chronic psoriasis for at least 6 months prior to randomization
* At least 10% Body Surface Area (BSA) of Psoriasis at screening and at randomization
* Static Physician Global Assessment (sPGA) score of at least 3 and Psoriasis Area and Severity Index (PASI) score of at least 12 at screening and at randomization
* Candidate for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Pustular, erythrodermic, and/or guttate forms of psoriasis
* History of drug-induced psoriasis
* Prior use of etanercept
* Clinically significant flare of psoriasis during the 12 weeks prior to randomization
* Concurrent or recent use of any biologic agent
* Received non-biologic systemic psoriasis therapy or phototherapy (including psoralens and ultraviolet A [PUVA], ultraviolet B [UVB]) within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to randomization
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to randomization and during the study
* Have participated in any study with interleukin 17 (IL-17) antagonists, including ixekizumab
* Serious disorder or illness other than plaque psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1346 (Actual)
Dates: Start 2012-07-28 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (100):
- United States (41):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bell Gardens, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oceanside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edgewater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ormond Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skokie, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Henderson, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newington, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Windsor, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., High Point, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hazleton, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Jordan, Utah
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autónoma de Buenosaire
- Bulgaria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varna
- Canada (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brampton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond Hill, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Windsor, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Drummondville, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago, Chile
- Germany (23):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ergolding
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freising
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friedrichshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mahlow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mönchengladbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northeim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schwerin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Hungary (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kecskemét
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Makó
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orosháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szombathely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey, Mexico
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krasnodar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolensk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

REFERENCES:
- [Derived] Egeberg A, Hawkes JE, Somani N, Burge R, See K, Gallo G, McKean-Matthews M, Gooderham M, Han G, Armstrong A. Sustained Improvements in Clinical and Patient-Reported Outcomes and Quality of Life Through 5 Years Among Ixekizumab-Treated Patients with Complete Clearance of Scalp Psoriasis by Week 60. Dermatol Ther (Heidelb). 2024 Apr;14(4):1007-1018. doi: 10.1007/s13555-024-01147-7. Epub 2024 Apr 22. PMID 38647975
- [Derived] Armstrong A, Gonzalez-Cantero A, Khattri S, Muzy G, Malatestinic WN, Lampropoulou A, Feely M, See SK, Mert C, Blauvelt A. Comparing Achievement of National Psoriasis Foundation Treatment Targets among Patients with Plaque Psoriasis Treated with Ixekizumab versus Other Biologics in Clinical and Real-World Studies. Dermatol Ther (Heidelb). 2024 Apr;14(4):933-952. doi: 10.1007/s13555-024-01136-w. Epub 2024 Mar 23. PMID 38521874
- [Derived] Kirkham BW, Egeberg A, Behrens F, Pinter A, Merola JF, Holzkamper T, Gallo G, Ng KJ, Bolce R, Schuster C, Nash P, Puig L. A Comprehensive Review of Ixekizumab Efficacy in Nail Psoriasis from Clinical Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Rheumatol Ther. 2023 Oct;10(5):1127-1146. doi: 10.1007/s40744-023-00553-1. Epub 2023 Jul 3. PMID 37400681
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Blauvelt A, Lebwohl MG, Mabuchi T, Leung A, Garrelts A, Crane H, ElMaraghy H, Patel H, Ridenour T, See K, Gallo G, Paul C. Long-term efficacy and safety of ixekizumab: A 5-year analysis of the UNCOVER-3 randomized controlled trial. J Am Acad Dermatol. 2021 Aug;85(2):360-368. doi: 10.1016/j.jaad.2020.11.022. Epub 2020 Nov 28. PMID 33253833
- [Derived] Rich P, Goldblum O, Disch D, Lin CY, Merola JF, Elewski B. Nail Psoriasis Does Not Affect Skin Response to Ixekizumab in Patients With Moderate-To-Severe Psoriasis. J Drugs Dermatol. 2020 Aug 1;19(8):741-746. doi: 10.36849/JDD.2020.5116. PMID 32845588
- [Derived] Yosipovitch G, Reich A, Steinhoff M, Beselin A, Kent T, Dossenbach M, Berggren L, Henneges C, Luger T. Impact of Ixekizumab Treatment on Itch and Psoriasis Area and Severity Index in Patients with Moderate-to-Severe Plaque Psoriasis: An Integrated Analysis of Two Phase III Randomized Studies. Dermatol Ther (Heidelb). 2018 Dec;8(4):621-637. doi: 10.1007/s13555-018-0267-9. Epub 2018 Nov 21. PMID 30465321
- [Derived] Reich K, Jackson K, Ball S, Garces S, Kerr L, Chua L, Muram TM, Blauvelt A. Ixekizumab Pharmacokinetics, Anti-Drug Antibodies, and Efficacy through 60 Weeks of Treatment of Moderate to Severe Plaque Psoriasis. J Invest Dermatol. 2018 Oct;138(10):2168-2173. doi: 10.1016/j.jid.2018.04.019. Epub 2018 May 8. PMID 29751001
- [Derived] Blauvelt A, Papp KA, Griffiths CEM, Puig L, Weisman J, Dutronc Y, Kerr LF, Ilo D, Mallbris L, Augustin M. Efficacy and Safety of Switching to Ixekizumab in Etanercept Non-Responders: A Subanalysis from Two Phase III Randomized Clinical Trials in Moderate-to-Severe Plaque Psoriasis (UNCOVER-2 and -3). Am J Clin Dermatol. 2017 Apr;18(2):273-280. doi: 10.1007/s40257-016-0246-9. PMID 28074446
- [Derived] van de Kerkhof P, Guenther L, Gottlieb AB, Sebastian M, Wu JJ, Foley P, Morita A, Goldblum O, Zhang L, Erickson J, Ball S, Rich P. Ixekizumab treatment improves fingernail psoriasis in patients with moderate-to-severe psoriasis: results from the randomized, controlled and open-label phases of UNCOVER-3. J Eur Acad Dermatol Venereol. 2017 Mar;31(3):477-482. doi: 10.1111/jdv.14033. Epub 2016 Dec 2. PMID 27910156
- [Derived] Gordon KB, Blauvelt A, Papp KA, Langley RG, Luger T, Ohtsuki M, Reich K, Amato D, Ball SG, Braun DK, Cameron GS, Erickson J, Konrad RJ, Muram TM, Nickoloff BJ, Osuntokun OO, Secrest RJ, Zhao F, Mallbris L, Leonardi CL; UNCOVER-1 Study Group; UNCOVER-2 Study Group; UNCOVER-3 Study Group. Phase 3 Trials of Ixekizumab in Moderate-to-Severe Plaque Psoriasis. N Engl J Med. 2016 Jul 28;375(4):345-56. doi: 10.1056/NEJMoa1512711. Epub 2016 Jun 8. PMID 27299809
- [Derived] Armstrong AW, Lynde CW, McBride SR, Stahle M, Edson-Heredia E, Zhu B, Amato D, Nikai E, Yang FE, Gordon KB. Effect of Ixekizumab Treatment on Work Productivity for Patients With Moderate-to-Severe Plaque Psoriasis: Analysis of Results From 3 Randomized Phase 3 Clinical Trials. JAMA Dermatol. 2016 Jun 1;152(6):661-9. doi: 10.1001/jamadermatol.2016.0269. PMID 26953848
- [Derived] Griffiths CE, Reich K, Lebwohl M, van de Kerkhof P, Paul C, Menter A, Cameron GS, Erickson J, Zhang L, Secrest RJ, Ball S, Braun DK, Osuntokun OO, Heffernan MP, Nickoloff BJ, Papp K; UNCOVER-2 and UNCOVER-3 investigators. Comparison of ixekizumab with etanercept or placebo in moderate-to-severe psoriasis (UNCOVER-2 and UNCOVER-3): results from two phase 3 randomised trials. Lancet. 2015 Aug 8;386(9993):541-51. doi: 10.1016/S0140-6736(15)60125-8. Epub 2015 Jun 10. PMID 26072109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study has 4 periods: Period 1 - Screening; Period 2 - Blinded Induction Dosing Period (Weeks 0 to 12); Period 3 - Long-Term Extension Period (Weeks 12 to 264); Period 4 - Post-Treatment Follow-Up Period (Minimum of 12 Weeks)
Groups:
- Placebo: Placebo (PBO) for ixekizumab (Week 0) given as 2 subcutaneous (SC) injections followed by placebo for ixekizumab Q2W (Weeks 2, 4, 6, 8, and 10). Placebo for etanercept (1 SC injection) given twice weekly (every 3-4 days) starting at Week 0 up to Week 12.
- 50 mg Etanercept (ETN): Etanercept 50 mg (1 SC injection) given twice weekly (every 3-4 days) starting at Week 0 and up to Week 12.
  Placebo for ixekizumab given as 2 SC injections (Week 0) followed by placebo for ixekizumab Q2W given as 1 SC injection (Weeks 2, 4, 6, 8, and 10).
- 80 mg Ixekizumab Dosing Regimen 2 (Q4W): A starting dose of 160 mg (Week 0) given as 2 SC injections followed by 80 mg given as 1 SC injection Q4W (Weeks 4 and 8). Placebo for ixekizumab given as 1 SC injection at Weeks 2, 6, and 10. Placebo for etanercept (1 SC injection) given twice weekly starting at Week 0 up to Week 12.
- 80 mg Ixekizumab Dosing Regimen 1 (Q2W): A starting dose of 160 mg (Week 0) given as 2 SC injections followed by 80 mg given as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
  Placebo for etanercept (1 SC injection) given twice weekly starting at Week 0 up to Week 12.
- PBO/IXE80Q4W: Participants who received placebo during the induction period and received 80 mg ixekizumab SC injection every four weeks (IXE80Q4W) in the Long-term extension period.
- ETN/IXE80Q4W: Participants who received Etanercept during the induction period and received IXE80Q4W in the long-term extension period.
- IXE80Q4W/IXE80Q4W: Participants who received 80 mg ixe Q4W during the induction period and received IXE80Q4W in the long-term extension period.
- IXE80Q2W/IXE80Q4W: Participants who received 80 mg ixe Q2W (IXE80Q2W) during the induction period and received IXE80Q4W in the long-term extension period.
- PBO Follow-Up Period: Participants who received PBO in the Induction Period and entered the Post-Treatment Follow-up Period.
- ETN Follow-Up Period: Participants who received etanercept (ETN) in the Induction Period and entered the Post-Treatment Follow-up Period.
- IXE80Q4W Follow-Up Period: Participants who received 80 mg ixe Q4W in the Induction Period and entered the Post-Treatment Follow-up Period.
- IXE80Q2W Follow-Up Period: Participants who received 80 mg ixe Q2W in the Induction Period and entered the Post-Treatment Follow-up Period.
Period: Blinded Induction Dosing (Week 0-12)
Arm/Group | Placebo | 50 mg Etanercept (ETN) | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) | PBO/IXE80Q4W | ETN/IXE80Q4W | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q4W | PBO Follow-Up Period | ETN Follow-Up Period | IXE80Q4W Follow-Up Period | IXE80Q2W Follow-Up Period
Started | 193 | 382 | 386 | 385 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 193 | 382 | 382 | 384 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 183 | 369 | 360 | 363 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 13 | 26 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 9 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 8 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Extension Period (Week 12-264)
Arm/Group | Placebo | 50 mg Etanercept (ETN) | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) | PBO/IXE80Q4W | ETN/IXE80Q4W | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q4W | PBO Follow-Up Period | ETN Follow-Up Period | IXE80Q4W Follow-Up Period | IXE80Q2W Follow-Up Period
Started | 0 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 0 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 0 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 0 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 183 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 369 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 360 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 362 (Participants completed prior period then proceeded to IXE80Q4W long-term extension period.) | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 183 | 369 | 360 | 362 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 135 | 256 | 244 | 255 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 48 | 113 | 116 | 107 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 16 | 34 | 43 | 30 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 11 | 30 | 29 | 27 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6 | 17 | 23 | 18 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 6 | 14 | 10 | 11 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 5 | 5 | 5 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Parent/Caregiver Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Missing Disposition Form | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Period: Follow-Up Period (Minimum of 12 Weeks)
Arm/Group | Placebo | 50 mg Etanercept (ETN) | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) | PBO/IXE80Q4W | ETN/IXE80Q4W | IXE80Q4W/IXE80Q4W | IXE80Q2W/IXE80Q4W | PBO Follow-Up Period | ETN Follow-Up Period | IXE80Q4W Follow-Up Period | IXE80Q2W Follow-Up Period
Started | 0 | 0 | 0 | 0 | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 157 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 309 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 305 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 313 (Participants who completed or discontinued from study treatment and entered the follow-up period.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 157 | 309 | 305 | 313
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 126 | 233 | 225 | 230
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 76 | 80 | 83
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 28 | 34 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 21 | 19 | 19
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 9 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9 | 8 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 4 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Placebo for ixekizumab (Week 0) given as 2 SC injections followed by placebo for ixekizumab Q2W (Weeks 2, 4, 6, 8, and 10). Placebo for etanercept (1 SC injection) given twice weekly (every 3-4 days) starting at Week 0 up to Week 12.
- 50 mg Etanercept: Etanercept 50 mg (1 SC injection) given twice weekly (every 3-4 days) starting at Week 0 and up to Week 12. Placebo for ixekizumab given as 2 SC injections (Week 0) followed by placebo for ixekizumab Q2W given as 1 SC injection (Weeks 2, 4, 6, 8, and 10).
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) | Total
Number analyzed (Participants) | 193 | 382 | 386 | 385 | 1346
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 180 | 349 | 358 | 351 | 1238
  >=65 years | 13 | 33 | 28 | 34 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 113 | 128 | 131 | 428
  Male | 137 | 269 | 258 | 254 | 918
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 52 | 50 | 57 | 184
  Not Hispanic or Latino | 133 | 263 | 269 | 259 | 924
  Unknown or Not Reported | 35 | 67 | 67 | 69 | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 4 | 1 | 10
  Asian | 7 | 11 | 11 | 12 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 4 | 6
  Black or African American | 8 | 10 | 9 | 5 | 32
  White | 176 | 351 | 360 | 361 | 1248
  More than one race | 1 | 5 | 1 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 2 | 7 | 6 | 6 | 21
  Chile | 11 | 21 | 22 | 22 | 76
  Mexico | 1 | 2 | 1 | 1 | 5
  Bulgaria | 9 | 12 | 14 | 13 | 48
  Germany | 45 | 87 | 90 | 90 | 312
  Hungary | 18 | 31 | 31 | 33 | 113
  Poland | 5 | 10 | 11 | 13 | 39
  Russia | 11 | 22 | 20 | 24 | 77
  Canada | 22 | 44 | 44 | 42 | 152
  United States | 69 | 146 | 147 | 141 | 503

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Static Physician Global Assessment (sPGA) of (0, 1) (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: sPGA)
Description: The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA (0,1) response was defined as a post-baseline sPGA score of 0 or 1.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet clinical response criteria or have missing data at Week 12 will be considered non-responders for the Non-Responder Imputation (NRI) analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 193 | 382 | 386 | 385
Participants | 13 | 159 | 291 | 310
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Number of Participants Achieving Psoriasis Area and Severity Index ≥75% (PASI 75) Improvement (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: PASI)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 was defined as having an improvement of at least 75% in the PASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 193 | 382 | 386 | 385
Participants | 14 | 204 | 325 | 336
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Participants Achieving an sPGA (0) (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: sPGA)
Description: The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA (0) response was defined as a post-baseline sPGA score of 0.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 193 | 382 | 386 | 385
Participants | 0 | 33 | 139 | 155
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants Achieving ≥90% (PASI 90) Improvement (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: PASI)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 90 were defined as having an improvement of at least 90% in the PASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 193 | 382 | 386 | 385
Participants | 6 | 98 | 252 | 262
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants Achieving 100% (PASI 100) Improvement (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: PASI)
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 100 were defined as having an improvement of at least 100% in the PASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 193 | 382 | 386 | 385
Participants | 0 | 28 | 135 | 145
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Number of Participants Achieving an Itch Numeric Rating Scale (NRS) ≥4 Point Reduction [Quality of Life and Outcome Assessments. Measures: Patient Reported Outcomes (PRO)]
Description: The Itch NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Participants indicate their overall severity of itching from Psoriasis by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Week 12
Population: All randomized participants and had an Itch NRS score >=4 at baseline. Participants who did not meet clinical response criteria or have missing data at Week 12 will be considered non-responders for the NRI analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 158 | 312 | 313 | 320
Participants | 33 | 200 | 250 | 264
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5 point change from baseline is considered clinically relevant. Least Square (LS) Means in total DLQI score were calculated using Mixed Model Repeated Measures (MMRM) with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants and had at least one post-dose measurement of DLQI.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 191 | 376 | 375 | 377
Units on a Scale | -1.7 (0.32) | -8.0 (0.23) | -9.6 (0.23) | -10.2 (0.23)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score
Description: The NAPSI is a numeric, reproducible, objective tool used to evaluate the severity of fingernail bed psoriasis and fingernail matrix psoriasis by area of involvement in the fingernail unit. The fingernail is divided with imaginary horizontal and longitudinal lines into quadrants. Each fingernail is given a score for fingernail bed psoriasis: 0 (none) to 4 (psoriasis in 4 quadrants of the nail) and fingernail matrix psoriasis (0 to 4) depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed and fingernail matrix psoriasis in each quadrant. The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). Each fingernail is evaluated, and the sum of all the fingernails is the total NAPSI score (range, 0 to 80). LS Means in NAPSI score were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants and had fingernail involvement at baseline and had at least one post-dose measurement of NAPSI.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 115 | 233 | 226 | 228
Units on a Scale | 1.6362 (1.0991) | -6.4015 (0.7716) | -9.9793 (0.7838) | -10.4145 (0.7820)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

9. Secondary Outcome: Percent of Body Surface Area (BSA) Involvement of Psoriasis
Description: Percentage involvement of psoriasis on each participants body surface area was assessed by the investigator on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand (including palm, fingers and thumb). LS Means in BSA were calculated using MMRM with baseline BSA as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Week 12
Population: All randomized participants and had at least one post-dose measurement of BSA.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 192 | 378 | 377 | 380
Percent | -0.7 (1.03) | -16.4 (0.73) | -23.2 (0.73) | -23.2 (0.73)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline in Psoriasis Scalp Severity Index (PSSI) Score
Description: PSSI is a composite score ranging from 0 (best) to 72 (worst), derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of scalp area involved. LS Means in PSSI score were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants and had scalp psoriasis at baseline and had at least one post-dose measurement of PSSI.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 175 | 345 | 344 | 344
Units on a Scale | -5.0 (0.53) | -15.9 (0.38) | -18.2 (0.38) | -18.8 (0.38)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

11. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Report 16 Items (QIDS-SR16) Total Score [Quality of Life and Outcome Assessments. Measures: Patient Reported Outcomes (PRO)]
Description: The QIDS-SR16 is a self-administered, 16-item instrument in which a participant is asked to consider each statement as it relates to the way they have felt for the past 7 days. There is a 4-point scale for each item ranging from 0 (best) to 3 (worst). The 16 items are scored to give 9 individual depression domains (sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance [initial, middle and late insomnia or hypersomnia], decrease/increase in appetite/weight, and psychomotor agitation/retardation), which are summed to give a single score ranging from 0 to 27, with higher scores denoting greater symptom severity. LS Means in total QIDS-SR16 score were calculated using the analysis of covariance (ANCOVA) model with treatment, pooled center and baseline QIDS total score.
Time Frame: Baseline, Week 12
Population: All randomized participants and had at least one post-dose measurement of QIDS-SR16. Participants with missing QIDS-SR16 data were imputed by Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 184 | 379 | 373 | 373
Units on a Scale | -0.3 (0.20) | -0.5 (0.14) | -0.9 (0.14) | -1.3 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p = 0.473, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p = 0.015, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, ANCOVA

12. Secondary Outcome: Change From Baseline in All Scores of the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO)
Description: The WPAI-PSO is a 6-item instrument used to assess the impact of psoriasis on productivity impairment within the past 7 days. It has four domains: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score, and impairment in daily activities performed outside of work. Four scores are derived as percentages: absenteeism, presenteeism, overall work impairment (absenteeism and presenteeism), and impairment in activities performed outside of work. Percentage is calculated as: each score * 100 and ranged from 0 to 100. Higher scores indicate greater impairment in productivity. LS Means in each WPAI-PSO score were calculated using the ANCOVA model with treatment, pooled center and baseline WPAI-PSO score.
Time Frame: Baseline, Week 12
Population: All randomized participants, even if the participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol, and had at least one post-dose measurement of WPAI-PSO. Participants with missing WPAI-PSO data were imputed by Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 184 | 376 | 375 | 373
Units on a Scale
  Absenteeism Score: number analyzed (Participants) | 120 | 217 | 230 | 218
  Absenteeism Score | 0.0 (0.82) | -2.8 (0.62) | -2.0 (0.60) | -2.5 (0.61)
  Activity Impairment Score | -2.5 (1.30) | -21.1 (0.91) | -23.3 (0.92) | -24.5 (0.92)
  Presenteeism Score: number analyzed (Participants) | 137 | 243 | 256 | 242
  Presenteeism Score | -0.8 (1.37) | -16.4 (1.04) | -16.0 (1.01) | -18.1 (1.04)
  Work Productively Loss Score: number analyzed (Participants) | 120 | 216 | 228 | 216
  Work Productively Loss Score | 0.6 (1.59) | -17.4 (1.20) | -16.7 (1.16) | -19.3 (1.19)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from Absenteeism Score; Test type: Superiority or Other; p = 0.006, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from Absenteeism Score; Test type: Superiority or Other; p = 0.045, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from Absenteeism Score; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from Work Productively Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 11: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from Work Productively Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from Work Productively Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA

13. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form (SF-36) Health Survey, Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. In this study, the SF-36 acute version was used, which has a 1 week recall period. LS Means in SF-36 score were calculated using the ANCOVA model with treatment, pooled center and baseline SF-36 score.
Time Frame: Baseline, Week 12
Population: All randomized participants and had at least one post-dose measurement of SF-36. Participants with missing SF-36 data were imputed by Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 179 | 365 | 362 | 357
Units on a Scale
  PCS | -0.1993 (0.5077) | 3.1176 (0.3568) | 4.1143 (0.3587) | 3.9620 (0.3604)
  MCS | 1.1305 (0.5768) | 2.6486 (0.4047) | 3.7961 (0.4074) | 4.2772 (0.4093)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from PCS; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from PCS; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from PCS; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs 50 mg Etanercept; Includes analysis only from MCS; Test type: Superiority or Other; p = 0.031, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Includes analysis only from MCS; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Includes analysis only from MCS; Test type: Superiority or Other; p < 0.001, ANCOVA

14. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Severity
Description: The Patient's Global Assessment of Disease Severity is a single-item participant-reported outcome measure on which participants are asked to rate the severity of their psoriasis "today" from 0 (Clear) = no psoriasis, to 5 (Severe) = the worst their psoriasis has ever been. LS Means in Patient's Global Assessment of Disease Severity score were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants and had at least one post-dose measurement of Patient's Global Assessment of Disease Severity.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 192 | 377 | 375 | 376
Units on a Scale | -0.5 (0.08) | -2.3 (0.06) | -3.1 (0.06) | -3.1 (0.06)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

15. Secondary Outcome: Number of Participants Achieving Palmoplantar PASI of ≥50% (PPASI 50) Improvement
Description: Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 to 72. Participants achieving PPASI 50 were defined as having an improvement of at least 50% in the PPASI scores compared to baseline.
Time Frame: Week 12
Population: All randomized participants and had a diagnosis of palmoplantar psoriasis at baseline. Participants who did not meet clinical response criteria or have missing data at Week 12 will be considered non-responders for the NRI analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 54 | 95 | 87 | 96
Participants | 26 | 77 | 75 | 78
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

16. Secondary Outcome: Number of Participants Achieving Palmoplantar PASI of ≥75% (PPASI 75) Improvement
Description: Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 to 72. Participants achieving PPASI 75 were defined as having an improvement of at least 75% in the PPASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 54 | 95 | 87 | 96
Participants | 19 | 63 | 69 | 72
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

17. Secondary Outcome: Number of Participants Achieving Palmoplantar PASI of 100% (PPASI 100) Improvement
Description: Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 to 72. Participants achieving PPASI 100 were defined as having an improvement of 100% in the PPASI scores compared to baseline.
Time Frame: Week 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 54 | 95 | 87 | 96
Participants | 15 | 57 | 54 | 61
Statistical Analysis 1: Comparison: Placebo vs 50 mg Etanercept; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 2 (Q4W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs 80 mg Ixekizumab Dosing Regimen 1 (Q2W); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

18. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Ixekizumab Antibodies
Description: The percentage of participants with treatment-emergent positive anti-ixekizumab antibodies at any time post-baseline were summarized by treatment group. Percentage of participants with treatment-emergent positive anti-ixekizumab antibodies were calculated as: number of participants with an evaluable baseline sample and ≥1 evaluable post-baseline sample/number of participants in the analysis population * 100.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study treatment and had evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W)
Number analyzed (Participants) | 191 | 378 | 378 | 378
Participants | 2 | 8 | 52 | 23

ADVERSE EVENTS:
Time Frame: Up to 288 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo: Placebo for ixekizumab administered by two SC injections at Week 0, then one SC injection per Dosing Regimen 1 (Q2W) until Week 12. Placebo for etanercept administered by one SC injection twice weekly starting at Week 0 up to Week 12. At Week 12, arm is assigned to Dosing Regimen 2 (Q4W).
- PBO/IXE80Q4W Long-Term Extension: Participants who received placebo during the induction period and received 80 mg ixekizumab SC injection every four weeks (IXE80Q4W) in the Long-term extension period.
- ETN/IXE80Q4W Long-Term Extension: Participants who received Etanercept during the induction period and received IXE80Q4W in the long-term extension period.
- IXE80Q4W/IXE80Q4W Long-Term Extension: Participants who received 80 mg ixe Q4W during the induction period and received IXE80Q4W in the long-term extension period.
- IXE80Q2W/IXE80Q4W Long-Term Extension: Participants who received 80 mg ixe Q2W (IXE80Q2W) during the induction period and received IXE80Q4W in the long-term extension period.
- ETN Follow-Up Period: Participants who received ETN in the Induction Period and entered the Post-Treatment Follow-up Period.
- IXE80Q4W Follow-Up: Participants who received 80 mg ixe Q4W in the Induction Period and entered the Post-Treatment Follow-up Period.
- IXE80Q2W Follow-Up: Participants who received 80 mg ixe Q2W in the Induction Period and entered the Post-Treatment Follow-up Period.
Arm/Group | Placebo | 50 mg Etanercept | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) | PBO/IXE80Q4W Long-Term Extension | ETN/IXE80Q4W Long-Term Extension | IXE80Q4W/IXE80Q4W Long-Term Extension | IXE80Q2W/IXE80Q4W Long-Term Extension | PBO Follow-Up Period | ETN Follow-Up Period | IXE80Q4W Follow-Up | IXE80Q2W Follow-Up
Serious Adverse Events (participants affected / at risk) | 5/193 | 8/382 | 6/382 | 9/384 | 45/183 | 71/369 | 82/360 | 55/362 | 5/157 | 5/309 | 2/305 | 6/313
Other Adverse Events (participants affected / at risk) | 40/193 | 90/382 | 115/382 | 123/384 | 117/183 | 240/369 | 236/360 | 249/362 | 9/157 | 23/309 | 14/305 | 15/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=193) | 50 mg Etanercept (N=382) | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) (N=382) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) (N=384) | PBO/IXE80Q4W Long-Term Extension (N=183) | ETN/IXE80Q4W Long-Term Extension (N=369) | IXE80Q4W/IXE80Q4W Long-Term Extension (N=360) | IXE80Q2W/IXE80Q4W Long-Term Extension (N=362) | PBO Follow-Up Period (N=157) | ETN Follow-Up Period (N=309) | IXE80Q4W Follow-Up (N=305) | IXE80Q2W Follow-Up (N=313)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gas gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0/137 (0) | 0/269 (0) | 0/254 (0) | 0/254 (0) | 0/129 (0) | 0/260 (0) | 1/241 (1) | 0/241 (0) | 0/108 (0) | 0/217 (0) | 0/205 (0) | 0/209 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biopsy liver (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (8) | 4 (7) | 4 (6) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ewing's sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease mixed cellularity stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 1/109 (1) | 0/119 (0) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/137 (0) | 0/269 (0) | 0/254 (0) | 0/254 (0) | 0/129 (0) | 1/260 (1) | 2/241 (2) | 2/241 (2) | 0/108 (0) | 0/217 (0) | 0/205 (0) | 0/209 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/137 (0) | 0/269 (0) | 0/254 (0) | 0/254 (0) | 0/129 (0) | 0/260 (0) | 1/241 (1) | 0/241 (0) | 0/108 (0) | 0/217 (0) | 0/205 (0) | 0/209 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/56 (0) | 1/113 (1) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 0/119 (0) | 1/121 (1) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Vulval cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 1/119 (1) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miller fisher syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 1/109 (1) | 2/119 (2) | 0/121 (0) | 0/49 (0) | 1/92 (1) | 0/100 (0) | 0/104 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 0/119 (0) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 1/100 (1) | 0/104 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar i disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/137 (0) | 0/269 (0) | 0/254 (0) | 0/254 (0) | 0/129 (0) | 1/260 (1) | 0/241 (0) | 0/241 (0) | 0/108 (0) | 0/217 (0) | 0/205 (0) | 0/209 (0)
Breast disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/56 (0) | 1/113 (1) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 0/119 (0) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Prostatitis (Reproductive system and breast disorders) | 0/137 (0) | 0/269 (0) | 1/254 (1) | 0/254 (0) | 0/129 (0) | 0/260 (0) | 0/241 (0) | 0/241 (0) | 0/108 (0) | 0/217 (0) | 0/205 (0) | 0/209 (0)
Uterine scar (Reproductive system and breast disorders) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 0/119 (0) | 1/121 (1) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 0/109 (0) | 1/119 (1) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Implantable cardiac monitor insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal operation (Surgical and medical procedures) | 0/56 (0) | 0/113 (0) | 0/128 (0) | 0/130 (0) | 0/54 (0) | 1/109 (1) | 0/119 (0) | 0/121 (0) | 0/49 (0) | 0/92 (0) | 0/100 (0) | 0/104 (0)
Air embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=193) | 50 mg Etanercept (N=382) | 80 mg Ixekizumab Dosing Regimen 2 (Q4W) (N=382) | 80 mg Ixekizumab Dosing Regimen 1 (Q2W) (N=384) | PBO/IXE80Q4W Long-Term Extension (N=183) | ETN/IXE80Q4W Long-Term Extension (N=369) | IXE80Q4W/IXE80Q4W Long-Term Extension (N=360) | IXE80Q2W/IXE80Q4W Long-Term Extension (N=362) | PBO Follow-Up Period (N=157) | ETN Follow-Up Period (N=309) | IXE80Q4W Follow-Up (N=305) | IXE80Q2W Follow-Up (N=313)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 3 (7) | 11 (12) | 10 (12) | 27 (29) | 14 (18) | 25 (32) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 3 (21) | 42 (207) | 43 (99) | 37 (111) | 18 (102) | 24 (186) | 34 (291) | 24 (169) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 6 (6) | 1 (1) | 17 (24) | 20 (23) | 24 (32) | 36 (47) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 12 (16) | 12 (13) | 5 (5) | 18 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 11 (16) | 20 (20) | 21 (23) | 20 (21) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (12) | 19 (22) | 29 (29) | 26 (31) | 55 (124) | 104 (196) | 107 (239) | 112 (222) | 4 (4) | 4 (4) | 5 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 7 (7) | 0 (0) | 4 (6) | 20 (26) | 17 (20) | 21 (23) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 16 (22) | 10 (11) | 28 (41) | 27 (47) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8) | 8 (8) | 8 (8) | 21 (27) | 33 (58) | 48 (67) | 42 (68) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 5 (5) | 5 (5) | 6 (9) | 18 (26) | 21 (25) | 21 (39) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/56 (1) | 1/113 (1) | 1/128 (1) | 1/130 (1) | 2/54 (3) | 2/109 (3) | 6/119 (13) | 4/121 (5) | 0/49 (0) | 0/92 (0) | 1/100 (1) | 0/104 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7) | 9 (9) | 13 (14) | 17 (17) | 20 (24) | 29 (38) | 41 (60) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 8 (8) | 7 (8) | 16 (19) | 28 (32) | 23 (33) | 30 (34) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (10) | 11 (15) | 16 (23) | 16 (20) | 9 (15) | 30 (47) | 23 (27) | 27 (39) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 9 (10) | 6 (6) | 11 (17) | 23 (29) | 14 (18) | 26 (29) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 6 (8) | 4 (4) | 10 (16) | 16 (16) | 14 (18) | 16 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 8 (9) | 7 (9) | 2 (2) | 20 (25) | 17 (22) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 5 (6) | 5 (5) | 12 (14) | 17 (22) | 17 (28) | 15 (17) | 3 (3) | 10 (10) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 9 (9) | 3 (3) | 5 (6) | 20 (24) | 30 (42) | 30 (31) | 26 (31) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days